CLINICAL TRIAL: NCT02676973
Title: Three Arm Apical Suspension Trial for Post-Hysterectomy Vault Prolapse: Prospective Randomized Trial Involving Sacral Colpopexy, Transvaginal Mesh and Native Tissue Apical Repair
Brief Title: Apical Suspension Repair for Vault Prolapse In a Three-Arm Randomized Trial Design
Acronym: ASPIRe
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: NICHD Pelvic Floor Disorders Network (Network)
Collaborators: The Cleveland Clinic (Other); University of Alabama at Birmingham (Other); University of California, San Diego (Other); Duke University (Other); University of New Mexico (Other); Women and Infants Hospital of Rhode Island (Other); RTI International (Other); University of Pennsylvania (Other); University of Pittsburgh (Other); Kaiser Permanente (Other); University of Texas Southwestern Medical Center (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 27P01; 1U01HD069031-01 (NIH); 2U10HD041261 (NIH); 2U10HD054215 (NIH); 2U10HD041267 (NIH); 1U10HD069006 (NIH); 2U10HD054214 (NIH); 1U10HD069013 (NIH); 1U10HD069025 (NIH); 1U10HD069010 (NIH); U10HD041263 (NIH)
Record Dates: First submitted 2015-11-30; First posted 2016-02-09 (Estimated); Results first posted 2024-05-17 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Visceral Prolapse
Keywords: pelvic organ prolapse; POP; vault prolapse; cystocele; vaginal prolapse; post-hysterectomy vaginal prolapse
MeSH Terms: conditions — Visceral Prolapse; Pelvic Organ Prolapse; Cystocele; Uterine Prolapse | interventions — Robotics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sacral Colpopexy (Active Comparator): Sacral Colpopexy performed via open, robotic, or laparoscopic procedure.
  Interventions: Procedure: Open, Robotic, or Laparoscopic
- Transvaginal Native Tissue Repair (Active Comparator): Transvaginal Native Tissue Repair: Sacrospinous Ligament Suspension (SSLS) and Uterosacral Ligament Suspension (USLS)
  Interventions: Procedure: Transvaginal Native Tissue Repair
- Apical Transvaginal Mesh Repair (Active Comparator): Uphold™ LITE
  Interventions: Procedure: Uphold™ LITE

INTERVENTIONS:
Procedure: Open, Robotic, or Laparoscopic — Sacral Colpopexy is a surgery performed either through an incision in the abdomen or through several small incisions with the help of a laparoscope (a slender tube) or robot. The surgery is done with a permanent synthetic (man-made) mesh. The mesh is sutured (stitched) to the vagina and sacrum (tail bone) and is used as reinforcement. It provides additional support to weakened tissues and/or muscles.
  Arms: Sacral Colpopexy
Procedure: Transvaginal Native Tissue Repair — Transvaginal Native Tissue Repair is a surgery performed with an incision through the vagina (transvaginal). The surgery is done using both permanent and absorbable sutures (stitches), to support weakened tissue and/or muscles, and attach the top of the vagina to ligaments in the pelvis (either to the sacrospinous ligament or uterosacral ligament).
  Arms: Transvaginal Native Tissue Repair
Procedure: Uphold™ LITE — Transvaginal Mesh Repair is a surgery performed with an incision through the vagina (transvaginal). The surgery is done with a permanent synthetic (man-made) mesh. The mesh is attached to ligaments in the pelvis and is used to reinforce natural tissue and/or muscles, which are no longer able to provide support to the vagina.
  Arms: Apical Transvaginal Mesh Repair

SUMMARY:
The study is a multi-center, randomized, surgical trial of women with symptomatic post-hysterectomy apical (cuff) prolapse desiring surgical treatment. This study will compare the three available surgical treatments performed in usual practice. The purpose of this study is to compare two commonly performed mesh apical repair (sacral colpopexy vs. Apical Transvaginal Mesh) and vaginal native tissue apical repairs with mesh reinforced repairs. The primary outcome is measured over time (up to 60 months) using a survival analysis approach. Participants will be followed for at least 36-months (3-years) post surgery and up to a maximum of 60-months (5-years) during the primary trial. Participants who complete the primary trial will be approached for consent for long-term follow-up as part of a study extension and will be followed up to a maximum of 120-months (10-years).

The investigators hypothesize that treatment failure will not differ between vaginally and abdominally placed mesh for vault vaginal prolapse, and mesh repairs (regardless of route of implantation) will be superior to native tissue apical suspension.

DETAILED DESCRIPTION:
The primary purpose of this three arm randomized clinical trial is to determine if apical transvaginal mesh placement is non-inferior to sacral colpopexy for anatomic correction of post-hysterectomy vaginal vault prolapse and to determine if mesh reinforced repairs performed by abdominal or vaginal approach are superior to native tissue vaginal repair. This trial has the following primary aims:

1. To determine if Apical Transvaginal Mesh is non-inferior to Sacral Colpopexy for anatomic correction of post-hysterectomy vaginal vault prolapse at time points through 3 years.

1A. In the case where Apical Transvaginal Mesh is shown to be statistically significantly non-inferior to Sacral Colpopexy for anatomic correction of post-hysterectomy vaginal vault prolapse at time points through 3 years, to determine if Apical Transvaginal Mesh is superior to Sacral Colpopexy for anatomic correction of post-hysterectomy vaginal vault prolapse at time points through 3 years.

2. To determine if Sacral Colpopexy is superior to Native Tissue Repair for anatomic correction of post-hysterectomy vaginal vault prolapse at time points through 3 years.

3. To determine if Apical Transvaginal Mesh is superior to Native Tissue Repair for anatomic correction of post-hysterectomy vaginal vault prolapse at time points through 3 years.

Additional secondary aims include:

1. Evaluate the development of a valid and reliable Global Composite Outcome that balances adverse events and patient-centered outcomes to anatomic definitions of failure and success.
2. Determine the impact of preoperative frailty and mobility on surgical treatment outcomes and postoperative complications of older women following surgical correction of apical pelvic organ prolapse.
3. Evaluate the patient's perspective about adverse events and their role in patient decision-making outcomes. The aims include comparing patient versus surgeon rankings of complication grade, outcome, expectedness and seriousness, to estimate the association between patient rankings of adverse events (AEs) with decision-making and quality of life outcomes and to determine if their perspective about AEs changes over time.

ELIGIBILITY:
Inclusion Criteria:

1. Women age 21 or older
2. Prior total hysterectomy (no cervix present)
3. Prolapse beyond the hymen (defined as Ba, C, or Bp > 0 cm)
4. Vaginal cuff descent into at least the lower two thirds of the vagina (defined as point C> -2/3 TVL)
5. Bothersome bulge symptoms as indicated on question 3 of the PFDI-20 form relating to 'sensation of bulging' or 'something falling out'
6. Desires surgical treatment for post-hysterectomy vaginal prolapse
7. Available for up to 60 month follow-up

Exclusion Criteria:

1. Previous synthetic material or biologic grafts (placed vaginally or abdominally) to augment POP repair including anterior, posterior and/or apical compartments
2. Known previous formal SSLS performed for either uterovaginal or post-hysterectomy vaginal vault prolapse *
3. Known adverse reaction to synthetic mesh or biological grafts; these complications include but are not limited to erosion, fistula, or abscess
4. Unresolved chronic pelvic pain-active
5. Prior abdominal or pelvic radiation
6. Contraindication to any of the index surgical procedures

   * Known Horseshoe Kidney or Pelvic Mass overlying the sacrum
   * Active diverticular abscess or active diverticulitis
   * Shortened vaginal length (<6 cm TVL)

     * NOTE:

       * Only documented SSLS will be an exclusion.
       * Mesh used for only mid-urethral sling will NOT be an exclusion
       * If prior POP repair is unknown and unable to be documented, subjects will be eligible based on clinician judgment. The investigator will examine and assess for evidence of mesh or graft if no evidence of mesh or graft is present on examination subject remains eligible.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 360 (Actual)
Dates: Start 2016-02-29 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2026-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Shawn Menefee, MD, Study Chair — Kaiser Permanente San Diego
Locations (10):
- United States (10):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California at San Diego, San Diego, California
  - Kaiser Permanente, San Diego, California
  - University of New Mexico, Albuquerque, New Mexico
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Brown/Women and Infants Hospital of Rhode Island, Providence, Rhode Island
  - University of Texas Southwestern Medical Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Menefee SA, Richter HE, Myers D, Moalli P, Weidner AC, Harvie HS, Rahn DD, Meriwether KV, Paraiso MFR, Whitworth R, Mazloomdoost D, Thomas S; NICHD Pelvic Floor Disorders Network. Apical Suspension Repair for Vaginal Vault Prolapse: A Randomized Clinical Trial. JAMA Surg. 2024 Aug 1;159(8):845-855. doi: 10.1001/jamasurg.2024.1206. PMID 38776067
- [Derived] Sung VW, Menefee S, Richter HE, Moalli PA, Andy U, Weidner A, Rahn DD, Paraiso MF, Jeney SE, Mazloomdoost D, Gilbert J, Whitworth R, Thomas S; Eunice Kennedy Shriver National Institute of Child Health and Human Development Pelvic Floor Disorders Network. Patient perspectives in adverse event reporting after vaginal apical prolapse surgery. Am J Obstet Gynecol. 2024 Aug;231(2):268.e1-268.e16. doi: 10.1016/j.ajog.2024.04.043. Epub 2024 May 6. PMID 38710268
- [Derived] Sung VW, Menefee S, Dunivan G, Richter HE, Moalli P, Weidner A, Andy UU, Jelovsek E, Mazloomdoost D, Whitworth R, Thomas S; NICHD Pelvic Floor Disorders Network. Design of a Study to Measure Patient-Perspectives in Adverse Event Reporting (the PPAR Study): Supplementary Study to the ASPIRe Trial. Female Pelvic Med Reconstr Surg. 2021 Jan 1;27(1):e112-e117. doi: 10.1097/SPV.0000000000000845. PMID 32487881
- [Derived] Menefee S, Richter HE, Myers D, Weidner A, Moalli P, Harvie H, Rahn D, Jeppson P, Paraiso M, Thomas S, Mazloomdoost D; NICHD Pelvic Floor Disorders Network. Design of a 3-Arm Randomized Trial for Posthysterectomy Vault Prolapse Involving Sacral Colpopexy, Transvaginal Mesh, and Native Tissue Apical Repair: The Apical Suspension Repair for Vault Prolapse in a Three-Arm Randomized Trial. Female Pelvic Med Reconstr Surg. 2020 Jul;26(7):415-424. doi: 10.1097/SPV.0000000000000803. PMID 31860566

RESULTS

PARTICIPANT FLOW:
Groups:
- Native Tissue: Transvaginal Native Tissue Repair: Transvaginal Native Tissue Repair is a surgery performed with an incision through the vagina (transvaginal). The surgery is done using both permanent and absorbable
- Sacral Colpopexy: Open, Robotic, or Laparoscopic: Sacral Colpopexy is a surgery performed either through an incision in the abdomen or through several small incisions with the help of a laparoscope (a slender tube) or
- Transvaginal Mesh: Uphold� LITE: Transvaginal Mesh Repair is a surgery performed with an incision through the vagina (transvaginal). The surgery is done with a permanent synthetic (man-made) mesh. The mesh is attached t
Period: Overall Study
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Started | 123 | 121 | 116
Completed | 104 | 100 | 92
Not Completed | 19 | 21 | 24
Not completed — Withdrawal by Subject | 9 | 8 | 11
Not completed — Lost to Follow-up | 8 | 12 | 8
Not completed — Death | 2 | 1 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh | Total
Number analyzed (Participants) | 123 | 121 | 116 | 360
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.4 (8.5) | 65.4 (8.6) | 66.4 (9.0) | 66.1 (8.7)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 123 | 121 | 116 | 360
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian/Alaskan Native | 5 | 1 | 0 | 6
  Asian | 1 | 1 | 1 | 3
  Black/African American | 10 | 13 | 12 | 35
  More than one race | 2 | 0 | 1 | 3
  Other | 4 | 4 | 3 | 11
  White | 101 | 102 | 99 | 302
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 15 | 12 | 48
  Not Hispanic or Latino | 98 | 103 | 104 | 305
  Unknown/ Not Reported | 4 | 3 | 0 | 7
Marital Status [Count of Participants; unit: Participants]
  Divorced/ Separated | 26 | 21 | 12 | 59
  MARRIED, HUSBAND IN LOUISIANA | 0 | 1 | 0 | 1
  Married /Living with partner | 82 | 77 | 85 | 244
  Single (never been married) | 7 | 8 | 4 | 19
  Widowed | 8 | 14 | 15 | 37
Education [Count of Participants; unit: Participants]
  4-Year College Degree | 24 | 23 | 23 | 70
  Associate College Degree | 28 | 34 | 35 | 97
  Graduate Degree | 11 | 12 | 5 | 28
  High School/GED | 47 | 39 | 40 | 126
  Less than High School | 10 | 9 | 11 | 30
  Unknown/ Not Reported | 3 | 4 | 2 | 9
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 27.9 (5.5) | 29.5 (6.4) | 28.7 (5.1) | 28.7 (5.8)
Current Smoker [Count of Participants; unit: Participants]
  No | 90 | 92 | 78 | 260
  Unknown | 25 | 22 | 27 | 74
  Yes | 8 | 7 | 11 | 26
Pregnancies [Median (Full Range); unit: Number of pregnancies] | 3 [1 to 9] | 3 [1 to 8] | 3 [1 to 7] | 3 [1 to 9]
Vaginal Deliveries [Median (Full Range); unit: Number of deliveries] | 3 [0 to 6] | 2 [1 to 8] | 2.5 [0 to 7] | 2 [0 to 8]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Considered Failures
Description: Failure was defined as any of the following: retreatment for prolapse, any POP-Q measure beyond the hymen, or presence of bother on PFDI vaginal bulge question. Under the permanent failure state assumption, the number of participants shown at each visit includes all participants who were still participating in the study or had a failure outcome prior their withdrawal. Similarly, the denominator number of participants for the cumulative failure at each visit includes all participants who were still participating in the study and attended the visit or had any failure outcome prior their withdrawal or missed visit.
Time Frame: 6 months through 60 Months
Population: An modified intent-to-treat (ITT) analysis which included all eligible participants who were randomized, received the randomized procedure, and who provided outcome data after baseline was performed.
Measure: Count of Participants; unit: Participants
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 118 | 120 | 113
Participants
  06 Months: number analyzed (Participants) | 112 | 114 | 111
  06 Months: Failure | 19 | 6 | 11
  06 Months: Non-failure | 93 | 108 | 100
  12 Months: number analyzed (Participants) | 112 | 109 | 107
  12 Months: Failure | 31 | 13 | 18
  12 Months: Non-failure | 81 | 96 | 89
  18 Months: number analyzed (Participants) | 106 | 104 | 103
  18 Months: Failure | 38 | 18 | 19
  18 Months: Non-failure | 68 | 86 | 84
  24 Months: number analyzed (Participants) | 105 | 104 | 107
  24 Months: Failure | 43 | 21 | 27
  24 Months: Non-failure | 62 | 83 | 80
  30 Months: number analyzed (Participants) | 102 | 99 | 105
  30 Months: Failure | 49 | 24 | 30
  30 Months: Non-failure | 53 | 75 | 75
  36 Months: number analyzed (Participants) | 106 | 100 | 100
  36 Months: Failure | 53 | 31 | 30
  36 Months: Non-failure | 53 | 69 | 70
  42 Months: number analyzed (Participants) | 95 | 90 | 93
  42 Months: Failure | 55 | 33 | 31
  42 Months: Non-failure | 40 | 57 | 62
  48 Months: number analyzed (Participants) | 93 | 86 | 84
  48 Months: Failure | 55 | 36 | 31
  48 Months: Non-failure | 38 | 50 | 53
  54 Months: number analyzed (Participants) | 84 | 66 | 74
  54 Months: Failure | 55 | 36 | 35
  54 Months: Non-failure | 29 | 30 | 39
  60 Months: number analyzed (Participants) | 76 | 63 | 60
  60 Months: Failure | 55 | 38 | 37
  60 Months: Non-failure | 21 | 25 | 23

2. Other Pre Specified Outcome: Change From Baseline PFDI Score
Description: The Pelvic Floor Distress Inventory is a 20-question, validated, self-reported instrument used to evaluate pelvic floor symptoms. It consists of an overall scale (range: 0-300) comprised of 3 sub-scales: 1. Pelvic Organ Prolapse Distress Inventory (range: 0-100), 2. Colorectal Anal Distress Inventory (range: 0-100), and 3. Urinary Distress Inventory (range: 0-100). The range of responses for all questions is 1-4 with (1) Not at all, (2) Somewhat, (3) Moderately, and (4), Quite a bit. Subscale scores are calculated by multiplying the mean value of all questions answered by 25 for the subscale. The range of score for each subscale is: 0-100 with 0 (least distress) to 100 (most distress). The PFDI is calculated as the sum of the three subscales. Lower scores indicate better function / fewer symptoms for the PFDI scale, POPDI subscale, CRADI subscale, and UDI subscale. Change from baseline = (Month [12, 24, 36] Score - Baseline Score).
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 117 | 120 | 113
units on a scale
  06 Months: number analyzed (Participants) | 112 | 114 | 111
  06 Months | -75.8 [-85.10 to -66.50] | -80.2 [-91.10 to -69.20] | -79.6 [-91.30 to -68.00]
  12 Months: number analyzed (Participants) | 111 | 109 | 104
  12 Months | -79.7 [-89.00 to -70.40] | -85.6 [-96.80 to -74.40] | -79.4 [-90.70 to -68.10]
  18 Months: number analyzed (Participants) | 102 | 102 | 101
  18 Months | -111.7 [-122.90 to -100.60] | -111.8 [-123.60 to -100.00] | -109 [-121.70 to -96.40]
  24 Months: number analyzed (Participants) | 97 | 97 | 105
  24 Months | -79.8 [-90.40 to -69.20] | -84.9 [-96.90 to -72.90] | -79.9 [-90.30 to -69.50]
  30 Months: number analyzed (Participants) | 91 | 95 | 100
  30 Months | -106.7 [-117.80 to -95.60] | -112 [-124.50 to -99.50] | -103.8 [-116.60 to -90.90]
  36 Months: number analyzed (Participants) | 94 | 94 | 93
  36 Months | -78.1 [-89.10 to -67.10] | -83.9 [-96.20 to -71.50] | -79.7 [-91.00 to -68.40]
  42 Months: number analyzed (Participants) | 77 | 83 | 82
  42 Months | -102.4 [-114.40 to -90.30] | -114.6 [-128.40 to -100.80] | -103.2 [-116.10 to -90.40]
  48 Months: number analyzed (Participants) | 76 | 73 | 74
  48 Months | -75.8 [-87.80 to -63.80] | -78.4 [-92.60 to -64.10] | -73.9 [-88.90 to -58.80]
  54 Months: number analyzed (Participants) | 58 | 45 | 53
  54 Months | -109.9 [-124.90 to -95.00] | -109.5 [-127.70 to -91.30] | -107 [-122.80 to -91.20]
  60 Months: number analyzed (Participants) | 41 | 37 | 37
  60 Months | -68.7 [-86.00 to -51.30] | -84.1 [-101.20 to -67.10] | -67.5 [-87.80 to -47.30]

3. Other Pre Specified Outcome: Change From Baseline CRADI Score
Description: as for outcome 2
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 116 | 118 | 112
units on a scale
  06 Months: number analyzed (Participants) | 112 | 114 | 111
  06 Months | -12.3 [-15.70 to -8.90] | -13.1 [-16.80 to -9.40] | -14.2 [-18.00 to -10.30]
  12 Months: number analyzed (Participants) | 111 | 109 | 104
  12 Months | -12.9 [-16.30 to -9.40] | -14.6 [-18.50 to -10.70] | -14.2 [-17.80 to -10.50]
  24 Months: number analyzed (Participants) | 97 | 97 | 105
  24 Months | -12.8 [-16.70 to -9.00] | -14.8 [-18.90 to -10.60] | -14 [-17.50 to -10.60]
  36 Months: number analyzed (Participants) | 94 | 94 | 93
  36 Months | -11.9 [-16.20 to -7.60] | -14.3 [-18.70 to -9.90] | -13.5 [-17.60 to -9.30]
  48 Months: number analyzed (Participants) | 76 | 73 | 74
  48 Months | -12.3 [-16.90 to -7.80] | -12.2 [-17.10 to -7.30] | -12.7 [-18.10 to -7.20]
  60 Months: number analyzed (Participants) | 41 | 37 | 37
  60 Months | -7.8 [-13.20 to -2.40] | -10.5 [-17.00 to -4.10] | -13.1 [-19.70 to -6.40]

4. Other Pre Specified Outcome: Change From Baseline POPDI Score
Description: as for outcome 2
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 117 | 120 | 113
units on a scale
  06 Months: number analyzed (Participants) | 112 | 114 | 111
  06 Months | -36.3 [-40.40 to -32.10] | -38 [-42.10 to -33.90] | -37.2 [-41.50 to -33.00]
  12 Months: number analyzed (Participants) | 111 | 109 | 104
  12 Months | -37.3 [-41.60 to -33.00] | -39.8 [-44.20 to -35.40] | -38.4 [-42.60 to -34.20]
  18 Months: number analyzed (Participants) | 102 | 102 | 101
  18 Months | -40.9 [-46.10 to -35.60] | -44.2 [-48.70 to -39.60] | -41.8 [-47.00 to -36.60]
  24 Months: number analyzed (Participants) | 97 | 97 | 105
  24 Months | -40.1 [-44.50 to -35.80] | -40.7 [-45.00 to -36.30] | -37.8 [-42.20 to -33.50]
  30 Months: number analyzed (Participants) | 91 | 95 | 100
  30 Months | -39.3 [-45.00 to -33.60] | -44.6 [-49.40 to -39.80] | -37.6 [-43.80 to -31.50]
  36 Months: number analyzed (Participants) | 94 | 94 | 93
  36 Months | -38.1 [-43.10 to -33.20] | -39.3 [-43.90 to -34.70] | -38.2 [-42.60 to -33.90]
  42 Months: number analyzed (Participants) | 77 | 83 | 82
  42 Months | -36.8 [-42.80 to -30.90] | -45.3 [-50.80 to -39.80] | -40.3 [-45.80 to -34.80]
  48 Months: number analyzed (Participants) | 76 | 73 | 74
  48 Months | -36.6 [-41.80 to -31.40] | -38.2 [-42.90 to -33.50] | -37.1 [-42.40 to -31.80]
  54 Months: number analyzed (Participants) | 58 | 45 | 53
  54 Months | -40.9 [-48.20 to -33.50] | -46.5 [-52.80 to -40.10] | -39.8 [-46.30 to -33.30]
  60 Months: number analyzed (Participants) | 41 | 37 | 37
  60 Months | -33.6 [-41.90 to -25.30] | -42.2 [-49.10 to -35.40] | -32.2 [-40.40 to -24.00]

5. Other Pre Specified Outcome: Change From Baseline UDI Score
Description: as for outcome 2
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 116 | 118 | 112
units on a scale
  06 Months: number analyzed (Participants) | 112 | 113 | 111
  06 Months | -27.3 [-32.10 to -22.40] | -29.3 [-35.10 to -23.40] | -28.2 [-34.10 to -22.30]
  12 Months: number analyzed (Participants) | 111 | 109 | 104
  12 Months | -29.5 [-34.10 to -25.00] | -31.2 [-36.80 to -25.70] | -26.9 [-32.70 to -21.10]
  24 Months: number analyzed (Participants) | 97 | 97 | 105
  24 Months | -26.8 [-32.10 to -21.50] | -29.5 [-35.40 to -23.50] | -28 [-33.30 to -22.70]
  36 Months: number analyzed (Participants) | 94 | 94 | 93
  36 Months | -28 [-33.00 to -23.00] | -30.2 [-36.00 to -24.40] | -28 [-33.70 to -22.30]
  48 Months: number analyzed (Participants) | 76 | 73 | 74
  48 Months | -26.9 [-33.10 to -20.60] | -27.9 [-35.40 to -20.50] | -24.1 [-31.40 to -16.80]
  60 Months: number analyzed (Participants) | 41 | 37 | 37
  60 Months | -27.3 [-36.40 to -18.20] | -31.4 [-40.40 to -22.30] | -22.2 [-32.10 to -12.40]

6. Other Pre Specified Outcome: Change From Baseline PFIQ Score
Description: The Pelvic Floor Impact Questionnaire short form (PFIQ-7) measuring the impact of bladder, bowel, and vaginal symptoms on a woman's daily activities, relationships and emotions is composed of an overall score (range 0-300), 3 subscales (7 questions each): the Urinary Impact Questionnaire (UIQ; range 0-100), the Pelvic Organ Prolapse Impact Questionnaire (POPIQ; range 0-100), and the Colorectal-Anal Impact Questionnaire (CRAIQ; range 0-100). The range of responses on all questions is 0-3 with (0) Not at all ... (3), Quite a bit. Subscale scores are calculated by multiplying the mean value of all answered questions for a scale by 100 divided by 3. The range of scores for each subscale is: 0-100 with 0 (least negative impact) to 100 (most negative impact). The PFIQ is the sum of the three subscales. Lower scores indicate better function / fewer symptoms for the PFIQ score, UIQ score, POPIQ score, and CRAIQ score. Change = (Week [12, 24] Score - Baseline Score).
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 116 | 118 | 112
units on a scale
  06 Months: number analyzed (Participants) | 112 | 114 | 110
  06 Months | -43.9 [-54.20 to -33.50] | -46.6 [-56.80 to -36.50] | -47 [-58.40 to -35.50]
  12 Months: number analyzed (Participants) | 110 | 109 | 104
  12 Months | -45.8 [-57.40 to -34.30] | -46.9 [-57.10 to -36.70] | -46.8 [-59.60 to -34.10]
  24 Months: number analyzed (Participants) | 97 | 97 | 105
  24 Months | -41.1 [-53.10 to -29.00] | -46.4 [-57.40 to -35.50] | -45.4 [-56.90 to -33.90]
  36 Months: number analyzed (Participants) | 93 | 93 | 93
  36 Months | -46.2 [-57.90 to -34.40] | -45.9 [-57.30 to -34.50] | -40.3 [-52.60 to -28.10]
  48 Months: number analyzed (Participants) | 75 | 73 | 74
  48 Months | -39.2 [-50.70 to -27.60] | -42.5 [-57.20 to -27.70] | -32.2 [-46.70 to -17.80]
  60 Months: number analyzed (Participants) | 41 | 37 | 37
  60 Months | -32.4 [-54.00 to -10.80] | -46.9 [-66.70 to -27.10] | -21.8 [-37.60 to -5.90]

7. Other Pre Specified Outcome: Change From Baseline CRAIQ Score
Description: as for outcome 6
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 115 | 118 | 112
units on a scale
  06 Months: number analyzed (Participants) | 111 | 113 | 109
  06 Months | -10.1 [-13.80 to -6.50] | -9.1 [-12.00 to -6.10] | -9.2 [-12.90 to -5.50]
  12 Months: number analyzed (Participants) | 110 | 108 | 102
  12 Months | -10.2 [-14.30 to -6.10] | -9.4 [-12.50 to -6.30] | -9.7 [-14.10 to -5.30]
  24 Months: number analyzed (Participants) | 97 | 96 | 105
  24 Months | -7.1 [-11.50 to -2.70] | -9.8 [-13.40 to -6.10] | -9.2 [-13.10 to -5.40]
  36 Months: number analyzed (Participants) | 93 | 93 | 92
  36 Months | -7.6 [-11.50 to -3.80] | -9.4 [-13.00 to -5.80] | -6.3 [-10.50 to -2.10]
  48 Months: number analyzed (Participants) | 74 | 73 | 74
  48 Months | -5.2 [-9.50 to -0.90] | -9.3 [-14.10 to -4.40] | -4.3 [-9.30 to 0.80]
  60 Months: number analyzed (Participants) | 41 | 37 | 37
  60 Months | -3.8 [-11.40 to 3.80] | -6.8 [-13.10 to -0.50] | -2.4 [-9.40 to 4.50]

8. Other Pre Specified Outcome: Change From Baseline POPIQ Score
Description: as for outcome 6
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 115 | 118 | 112
units on a scale
  06 Months: number analyzed (Participants) | 111 | 113 | 109
  06 Months | -19 [-23.60 to -14.30] | -19 [-23.80 to -14.10] | -19.1 [-23.80 to -14.30]
  12 Months: number analyzed (Participants) | 110 | 108 | 102
  12 Months | -18.6 [-23.40 to -13.80] | -19.5 [-24.10 to -14.90] | -18.2 [-23.40 to -13.00]
  24 Months: number analyzed (Participants) | 97 | 96 | 105
  24 Months | -18.3 [-23.50 to -13.10] | -20 [-24.50 to -15.50] | -18.4 [-23.20 to -13.60]
  36 Months: number analyzed (Participants) | 93 | 93 | 92
  36 Months | -20.9 [-26.20 to -15.60] | -18.8 [-23.50 to -14.10] | -17.9 [-22.60 to -13.10]
  48 Months: number analyzed (Participants) | 73 | 73 | 74
  48 Months | -17.9 [-24.10 to -11.70] | -17.3 [-23.20 to -11.40] | -17 [-22.80 to -11.20]
  60 Months: number analyzed (Participants) | 41 | 37 | 37
  60 Months | -17.1 [-26.80 to -7.30] | -22.3 [-31.30 to -13.30] | -10.9 [-16.90 to -4.90]

9. Other Pre Specified Outcome: Change From Baseline UIQ Score
Description: as for outcome 6
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 116 | 118 | 112
units on a scale
  06 Months: number analyzed (Participants) | 112 | 114 | 110
  06 Months | -15 [-19.40 to -10.60] | -18.7 [-23.40 to -14.10] | -18.9 [-23.90 to -13.90]
  12 Months: number analyzed (Participants) | 110 | 109 | 104
  12 Months | -17 [-21.50 to -12.60] | -18.3 [-22.80 to -13.80] | -18.5 [-23.20 to -13.70]
  24 Months: number analyzed (Participants) | 97 | 97 | 105
  24 Months | -15.7 [-20.30 to -11.00] | -17 [-22.00 to -11.90] | -17.8 [-22.50 to -13.00]
  36 Months: number analyzed (Participants) | 93 | 93 | 93
  36 Months | -17.6 [-22.70 to -12.60] | -17.7 [-22.90 to -12.50] | -16.3 [-21.60 to -11.00]
  48 Months: number analyzed (Participants) | 75 | 73 | 74
  48 Months | -16.3 [-21.20 to -11.30] | -15.9 [-22.00 to -9.90] | -11 [-16.90 to -5.00]
  60 Months: number analyzed (Participants) | 41 | 37 | 37
  60 Months | -11.5 [-19.70 to -3.30] | -17.8 [-26.30 to -9.20] | -8.4 [-14.70 to -2.00]

10. Other Pre Specified Outcome: Change From Baseline Functional Activity Scale
Description: Functional Activity Scale measuring the impact of incontinence symptoms on a woman's daily activities is composed of 13 questions about normal and physically strenuous daily activities. The range of responses on the individual questions is (1) No difficulty,... (5) Not able to do it. Scores are calculated by subtracting from the maximum sum (5*13=65) the product of the mean response and number of questions, then dividing by the total range of sums (65 - 13 = 52) and multiplying by 100. The range of responses is: 0-100 with 0 (worse functionality) to 100 (Better functionality). Change = (Month [6, 12, 18, 24, and 36] Score - Baseline Score).
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 116 | 117 | 112
units on a scale
  06 Months: number analyzed (Participants) | 112 | 113 | 110
  06 Months | 3.9 [1.60 to 6.20] | 6.2 [3.10 to 9.30] | 6.6 [3.50 to 9.70]
  12 Months: number analyzed (Participants) | 111 | 105 | 104
  12 Months | 4.6 [2.20 to 7.00] | 5.3 [2.20 to 8.40] | 6.1 [3.00 to 9.30]
  24 Months: number analyzed (Participants) | 96 | 96 | 105
  24 Months | 3.5 [0.60 to 6.50] | 6.1 [2.70 to 9.50] | 5.7 [2.70 to 8.70]
  36 Months: number analyzed (Participants) | 94 | 93 | 90
  36 Months | 2.6 [-0.40 to 5.50] | 7 [3.50 to 10.40] | 4.9 [1.50 to 8.30]
  48 Months: number analyzed (Participants) | 76 | 72 | 73
  48 Months | 2.4 [-1.50 to 6.40] | 5.3 [1.90 to 8.70] | 2.7 [-1.30 to 6.60]
  60 Months: number analyzed (Participants) | 41 | 37 | 35
  60 Months | -0.8 [-3.80 to 2.10] | 7.3 [2.20 to 12.30] | -0.7 [-5.20 to 3.90]

11. Other Pre Specified Outcome: Change From Baseline Body Part Pain Scale
Description: The Body Part Pain Scale measuring the pain experienced in the lower abdomen and pelvic region of the body is composed of 7 questions, each with a yes (1) or no (0) questions about experiencing pain followed by an intensity rating: 0 (No pain),..., 10 (Most intense). The score is calculated as the average of the responses. The range of responses is: 0-10 with 0 (No pain) to 10 (most intense pain). Lower scores indicate better function / fewer symptoms. Change = (Month [6, 12, 18, 24, and 36] Score - Baseline Score).
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 116 | 117 | 112
units on a scale
  06 Months: number analyzed (Participants) | 111 | 113 | 111
  06 Months | -0.4 [-0.60 to -0.10] | -0.5 [-0.70 to -0.20] | -0.6 [-0.90 to -0.40]
  12 Months: number analyzed (Participants) | 111 | 108 | 104
  12 Months | -0.4 [-0.60 to -0.20] | -0.5 [-0.70 to -0.20] | -0.7 [-1.00 to -0.40]
  24 Months: number analyzed (Participants) | 97 | 96 | 104
  24 Months | -0.4 [-0.70 to -0.20] | -0.5 [-0.80 to -0.20] | -0.7 [-0.90 to -0.40]
  36 Months: number analyzed (Participants) | 94 | 93 | 93
  36 Months | -0.3 [-0.50 to -0.10] | -0.6 [-0.90 to -0.20] | -0.7 [-1.00 to -0.40]
  48 Months: number analyzed (Participants) | 76 | 73 | 74
  48 Months | -0.2 [-0.40 to 0.00] | -0.5 [-0.80 to -0.10] | -0.5 [-0.70 to -0.20]
  60 Months: number analyzed (Participants) | 41 | 37 | 37
  60 Months | -0.3 [-0.50 to 0.00] | -0.7 [-1.10 to -0.30] | -0.2 [-0.60 to 0.20]

12. Other Pre Specified Outcome: Change From Baseline Surgical Pain Scale Rest Score
Description: The Surgical Pain Scale measuring the post-surgical pain experienced by a subject is composed of 4 questions: Pain at Rest (range 0-10), Pain with Normal Activities (range 0-10), Pain with Exercise (range 0-10), and Intensity of Worst Pain (range 0-10). Lower scores indicate better less pain for the Rest subscale, Normal subscale, Exercise Subscale, and Worst Subscale. Change = (Month [6, 12, 18, 24, and 36] Score - Baseline Score).
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 116 | 118 | 112
units on a scale
  06 Months: number analyzed (Participants) | 112 | 114 | 111
  06 Months | -0.6 [-1.00 to -0.20] | -0.5 [-0.90 to -0.10] | -0.7 [-1.10 to -0.30]
  12 Months: number analyzed (Participants) | 111 | 108 | 104
  12 Months | -0.5 [-1.00 to -0.10] | -0.4 [-0.80 to 0.10] | -0.8 [-1.20 to -0.40]
  24 Months: number analyzed (Participants) | 97 | 97 | 104
  24 Months | -0.5 [-1.00 to 0.00] | -0.4 [-0.90 to 0.10] | -0.6 [-1.10 to -0.20]
  36 Months: number analyzed (Participants) | 94 | 94 | 93
  36 Months | -0.5 [-0.90 to 0.00] | -0.6 [-1.10 to -0.20] | -0.2 [-0.70 to 0.30]
  48 Months: number analyzed (Participants) | 76 | 73 | 73
  48 Months | -0.9 [-1.40 to -0.40] | -0.5 [-1.00 to 0.10] | -0.2 [-0.80 to 0.50]
  60 Months: number analyzed (Participants) | 41 | 37 | 37
  60 Months | -0.7 [-1.50 to 0.00] | -1.1 [-2.00 to -0.30] | 0.2 [-0.70 to 1.00]

13. Other Pre Specified Outcome: Change From Baseline Surgical Pain Scale Normal Score
Description: as for outcome 12
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 116 | 118 | 112
units on a scale
  06 Months: number analyzed (Participants) | 112 | 114 | 111
  06 Months | -0.5 [-0.90 to -0.10] | -0.7 [-1.20 to -0.20] | -0.9 [-1.40 to -0.40]
  12 Months: number analyzed (Participants) | 111 | 108 | 104
  12 Months | -0.5 [-0.90 to -0.10] | -0.5 [-1.00 to -0.10] | -1 [-1.50 to -0.50]
  24 Months: number analyzed (Participants) | 97 | 97 | 104
  24 Months | -0.6 [-1.00 to -0.20] | -0.8 [-1.30 to -0.30] | -1 [-1.50 to -0.40]
  36 Months: number analyzed (Participants) | 94 | 94 | 93
  36 Months | -0.5 [-1.00 to 0.10] | -0.7 [-1.20 to -0.20] | -0.5 [-1.00 to 0.10]
  48 Months: number analyzed (Participants) | 76 | 73 | 74
  48 Months | -0.4 [-1.10 to 0.20] | -0.6 [-1.10 to 0.00] | -0.6 [-1.30 to 0.10]
  60 Months: number analyzed (Participants) | 41 | 37 | 37
  60 Months | -0.4 [-1.10 to 0.30] | -1 [-2.00 to 0.00] | 0.5 [-0.70 to 1.60]

14. Other Pre Specified Outcome: Change From Baseline Surgical Pain Scale Exercise Score
Description: as for outcome 12
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 75 | 74 | 74
units on a scale
  06 Months: number analyzed (Participants) | 51 | 51 | 56
  06 Months | -0.6 [-1.40 to 0.20] | -1.5 [-2.40 to -0.50] | -1.7 [-2.50 to -0.80]
  12 Months: number analyzed (Participants) | 57 | 49 | 51
  12 Months | -0.8 [-1.40 to -0.20] | -1.4 [-2.30 to -0.50] | -1.3 [-2.20 to -0.50]
  24 Months: number analyzed (Participants) | 48 | 39 | 50
  24 Months | -1.3 [-2.20 to -0.40] | -0.4 [-1.50 to 0.70] | -1.6 [-2.60 to -0.60]
  36 Months: number analyzed (Participants) | 42 | 42 | 41
  36 Months | -1.1 [-2.00 to -0.10] | -1.2 [-2.10 to -0.20] | -1.7 [-2.70 to -0.70]
  48 Months: number analyzed (Participants) | 33 | 35 | 29
  48 Months | -1.3 [-2.60 to -0.10] | -0.7 [-1.80 to 0.50] | -1.4 [-2.70 to 0.00]
  60 Months: number analyzed (Participants) | 21 | 21 | 9
  60 Months | -0.6 [-1.70 to 0.50] | -2.9 [-4.40 to -1.50] | 0.4 [-1.60 to 2.40]

15. Other Pre Specified Outcome: Change From Baseline Surgical Pain Scale Worst Score
Description: as for outcome 12
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 116 | 118 | 112
units on a scale
  06 Months: number analyzed (Participants) | 112 | 114 | 111
  06 Months | -0.7 [-1.10 to -0.20] | -1.1 [-1.70 to -0.50] | -0.9 [-1.40 to -0.40]
  12 Months: number analyzed (Participants) | 110 | 108 | 104
  12 Months | -0.8 [-1.20 to -0.40] | -0.9 [-1.50 to -0.40] | -1.1 [-1.60 to -0.60]
  24 Months: number analyzed (Participants) | 97 | 97 | 104
  24 Months | -0.6 [-1.20 to 0.00] | -1.2 [-1.80 to -0.60] | -1 [-1.50 to -0.50]
  36 Months: number analyzed (Participants) | 94 | 94 | 93
  36 Months | -0.4 [-1.00 to 0.20] | -1.1 [-1.80 to -0.50] | -0.4 [-1.00 to 0.10]
  48 Months: number analyzed (Participants) | 76 | 73 | 74
  48 Months | -0.3 [-1.00 to 0.50] | -1 [-1.60 to -0.30] | -0.2 [-0.80 to 0.40]
  60 Months: number analyzed (Participants) | 41 | 37 | 36
  60 Months | -0.6 [-1.30 to 0.20] | -1.7 [-2.70 to -0.70] | 0.8 [-0.10 to 1.60]

16. Other Pre Specified Outcome: Change From Baseline PISQ-IR Sexually Active Average Score
Description: The Pelvic Organ Prolapse Incontinence Sexual Questionnaire, IUGA-revised (PISQ-IR) is a questionnaire measuring the impact of incontinence symptoms on sexual function and satisfaction. The PISQ-IR Sexually Active-Average Score (SA-AVG) ranges from 0 to 5 with higher scores indicating better function/satisfaction. The change from baseline outcome is calculated as the difference in score at 6, 12, 18, 24, and 36 months and the score at baseline.
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 44 | 43 | 46
units on a scale
  06 Months: number analyzed (Participants) | 38 | 37 | 41
  06 Months | 0.4 [0.20 to 0.50] | 0.4 [0.20 to 0.60] | 0.5 [0.40 to 0.70]
  12 Months: number analyzed (Participants) | 36 | 36 | 40
  12 Months | 0.4 [0.20 to 0.60] | 0.4 [0.20 to 0.70] | 0.6 [0.50 to 0.80]
  24 Months: number analyzed (Participants) | 32 | 31 | 40
  24 Months | 0.4 [0.20 to 0.60] | 0.4 [0.20 to 0.70] | 0.5 [0.30 to 0.70]
  36 Months: number analyzed (Participants) | 28 | 30 | 34
  36 Months | 0.4 [0.10 to 0.60] | 0.4 [0.10 to 0.70] | 0.6 [0.40 to 0.80]
  48 Months: number analyzed (Participants) | 20 | 26 | 18
  48 Months | 0.3 [0.10 to 0.50] | 0.3 [0.10 to 0.60] | 0.4 [0.20 to 0.70]
  60 Months: number analyzed (Participants) | 10 | 14 | 12
  60 Months | 0.2 [0.00 to 0.50] | 0.6 [0.00 to 1.10] | 0.3 [0.00 to 0.70]

17. Other Pre Specified Outcome: Change From Baseline POP-Q Ba Measurement
Description: POPQ Point Ba represents the most distal (i.e. most dependent) position of any part of the upper anterior vaginal wall (between the vaginal cuff or anterior vaginal fornix and Point Aa). Point Ba coincides with Point Aa (-3 cm) in a woman who has no anterior POP. In a woman with severe POP, Ba coincides with Point C.
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 117 | 118 | 110
cm
  06 Months: number analyzed (Participants) | 112 | 114 | 110
  06 Months | -3.9 [-4.3 to -3.4] | -4.5 [-4.9 to -4.1] | -4.6 [-5.1 to -4.2]
  12 Months: number analyzed (Participants) | 106 | 105 | 103
  12 Months | -3.7 [-4.2 to -3.3] | -4.5 [-4.9 to -4.1] | -4.3 [-4.8 to -3.8]
  18 Months: number analyzed (Participants) | 94 | 94 | 92
  18 Months | -3.7 [-4.2 to -3.2] | -4.5 [-4.9 to -4.0] | -4.5 [-5.0 to -3.9]
  24 Months: number analyzed (Participants) | 88 | 86 | 96
  24 Months | -3.8 [-4.3 to -3.3] | -4.3 [-4.7 to -3.8] | -4.4 [-4.9 to -3.9]
  30 Months: number analyzed (Participants) | 77 | 81 | 80
  30 Months | -3.6 [-4.1 to -3.1] | -4.6 [-5.0 to -4.1] | -4.2 [-4.8 to -3.7]
  36 Months: number analyzed (Participants) | 84 | 78 | 82
  36 Months | -3.5 [-4.0 to -3.0] | -4.6 [-5.2 to -4.1] | -4.4 [-5.0 to -3.9]
  42 Months: number analyzed (Participants) | 53 | 66 | 66
  42 Months | -3.7 [-4.3 to -3.0] | -4.4 [-5.0 to -3.8] | -4.3 [-4.9 to -3.7]
  48 Months: number analyzed (Participants) | 56 | 52 | 62
  48 Months | -3.7 [-4.3 to -3.1] | -4.6 [-5.3 to -3.9] | -4.4 [-5.1 to -3.7]
  54 Months: number analyzed (Participants) | 41 | 35 | 41
  54 Months | -3.5 [-4.2 to -2.7] | -4.5 [-5.2 to -3.8] | -4.4 [-5.3 to -3.5]
  60 Months: number analyzed (Participants) | 34 | 34 | 35
  60 Months | -3.8 [-4.6 to -3.0] | -4.3 [-5.0 to -3.7] | -3.6 [-4.6 to -2.7]

18. Other Pre Specified Outcome: Change From Baseline POP-Q Bp Measurement
Description: POP-Q Point Bp represents the most distal position of any part of the upper posterior vaginal wall (between the vaginal cuff or posterior vaginal fornix and Point Ap).
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 117 | 118 | 110
cm
  06 Months: number analyzed (Participants) | 112 | 114 | 110
  06 Months | -2.6 [-3.2 to -2.0] | -2.8 [-3.3 to -2.2] | -3.2 [-3.7 to -2.6]
  12 Months: number analyzed (Participants) | 106 | 105 | 103
  12 Months | -2.6 [-3.2 to -2.0] | -2.9 [-3.5 to -2.3] | -3 [-3.5 to -2.4]
  18 Months: number analyzed (Participants) | 94 | 94 | 92
  18 Months | -2.4 [-3.0 to -1.7] | -2.8 [-3.5 to -2.2] | -3.1 [-3.8 to -2.4]
  24 Months: number analyzed (Participants) | 88 | 86 | 96
  24 Months | -2.5 [-3.2 to -1.9] | -2.5 [-3.1 to -1.8] | -2.9 [-3.5 to -2.2]
  30 Months: number analyzed (Participants) | 77 | 81 | 80
  30 Months | -2.8 [-3.5 to -2.1] | -2.5 [-3.2 to -1.9] | -2.8 [-3.5 to -2.1]
  36 Months: number analyzed (Participants) | 84 | 78 | 82
  36 Months | -2.3 [-3.0 to -1.7] | -2.5 [-3.2 to -1.8] | -2.8 [-3.5 to -2.2]
  42 Months: number analyzed (Participants) | 53 | 66 | 66
  42 Months | -2.1 [-2.9 to -1.3] | -2.8 [-3.5 to -2.0] | -3 [-3.8 to -2.3]
  48 Months: number analyzed (Participants) | 56 | 52 | 62
  48 Months | -2.6 [-3.5 to -1.8] | -2.6 [-3.4 to -1.8] | -3.4 [-4.2 to -2.6]
  54 Months: number analyzed (Participants) | 41 | 35 | 41
  54 Months | -2.7 [-3.7 to -1.7] | -2.5 [-3.5 to -1.5] | -3.1 [-4.0 to -2.2]
  60 Months: number analyzed (Participants) | 34 | 34 | 35
  60 Months | -2.6 [-3.8 to -1.5] | -2.3 [-3.3 to -1.3] | -3.1 [-4.1 to -2.1]

19. Other Pre Specified Outcome: Change From Baseline POP-Q C Measurement
Description: POP-Q Point C is measured in cm relative to the hymen with negative values being proximal to the hymen and positive values distal to the hymen. Point C represents either the most distal edge of the cervix or the leading edge of the vaginal cuff after total hysterectomy.
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 117 | 118 | 110
cm
  06 Months: number analyzed (Participants) | 112 | 114 | 110
  06 Months | -5.1 [-5.8 to -4.3] | -6.9 [-7.6 to -6.3] | -6.1 [-6.8 to -5.3]
  12 Months: number analyzed (Participants) | 106 | 105 | 103
  12 Months | -5.1 [-5.8 to -4.4] | -6.8 [-7.6 to -6.1] | -5.8 [-6.5 to -5.1]
  18 Months: number analyzed (Participants) | 94 | 94 | 92
  18 Months | -4.9 [-5.7 to -4.2] | -6.8 [-7.5 to -6.1] | -5.9 [-6.7 to -5.0]
  24 Months: number analyzed (Participants) | 88 | 86 | 96
  24 Months | -5 [-5.8 to -4.2] | -6.5 [-7.2 to -5.8] | -5.7 [-6.4 to -4.9]
  30 Months: number analyzed (Participants) | 77 | 81 | 80
  30 Months | -4.7 [-5.5 to -3.9] | -7.1 [-7.8 to -6.3] | -5.4 [-6.2 to -4.6]
  36 Months: number analyzed (Participants) | 84 | 78 | 82
  36 Months | -4.6 [-5.4 to -3.9] | -7.1 [-7.9 to -6.3] | -5.7 [-6.5 to -4.9]
  42 Months: number analyzed (Participants) | 53 | 66 | 66
  42 Months | -4.5 [-5.4 to -3.5] | -7 [-7.9 to -6.1] | -5.6 [-6.6 to -4.7]
  48 Months: number analyzed (Participants) | 56 | 52 | 62
  48 Months | -4.5 [-5.5 to -3.6] | -6.4 [-7.4 to -5.4] | -6.1 [-7.2 to -5.0]
  54 Months: number analyzed (Participants) | 41 | 35 | 41
  54 Months | -4.5 [-5.7 to -3.3] | -6.6 [-7.9 to -5.4] | -5.8 [-7.1 to -4.6]
  60 Months: number analyzed (Participants) | 34 | 34 | 35
  60 Months | -5.2 [-6.5 to -3.9] | -6.5 [-7.5 to -5.4] | -5.5 [-6.6 to -4.3]

20. Other Pre Specified Outcome: Change From Baseline POP-Q TVL Measurement
Description: POP-Q Total Vaginal Length (TVL) is measured in cm. It is the length of the vagina from posterior fornix to the hymen when Point C or D is reduced to its full normal position.
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 117 | 118 | 110
cm
  06 Months: number analyzed (Participants) | 112 | 114 | 110
  06 Months | -0.9 [-1.1 to -0.7] | 0.1 [-0.2 to 0.4] | -0.9 [-1.2 to -0.6]
  12 Months: number analyzed (Participants) | 106 | 105 | 103
  12 Months | -1 [-1.3 to -0.8] | 0 [-0.3 to 0.3] | -0.8 [-1.1 to -0.6]
  18 Months: number analyzed (Participants) | 94 | 94 | 92
  18 Months | -1.1 [-1.4 to -0.8] | 0 [-0.3 to 0.3] | -0.9 [-1.2 to -0.6]
  24 Months: number analyzed (Participants) | 88 | 86 | 96
  24 Months | -0.9 [-1.2 to -0.7] | 0 [-0.4 to 0.3] | -0.9 [-1.3 to -0.6]
  30 Months: number analyzed (Participants) | 77 | 81 | 80
  30 Months | -1.2 [-1.5 to -0.9] | 0.2 [-0.1 to 0.6] | -0.9 [-1.2 to -0.6]
  36 Months: number analyzed (Participants) | 84 | 78 | 82
  36 Months | -0.9 [-1.2 to -0.6] | 0.2 [-0.1 to 0.5] | -1 [-1.3 to -0.7]
  42 Months: number analyzed (Participants) | 53 | 66 | 66
  42 Months | -1 [-1.3 to -0.6] | -0.1 [-0.4 to 0.3] | -1.1 [-1.5 to -0.7]
  48 Months: number analyzed (Participants) | 56 | 52 | 62
  48 Months | -1.1 [-1.5 to -0.7] | 0 [-0.5 to 0.5] | -0.8 [-1.2 to -0.5]
  54 Months: number analyzed (Participants) | 41 | 35 | 41
  54 Months | -1 [-1.5 to -0.4] | -0.1 [-0.8 to 0.5] | -0.9 [-1.3 to -0.4]
  60 Months: number analyzed (Participants) | 34 | 34 | 35
  60 Months | -0.8 [-1.2 to -0.3] | -0.3 [-0.8 to 0.2] | -0.8 [-1.3 to -0.3]

21. Other Pre Specified Outcome: Number of Participants With PGI-I Reported Improvement
Description: The Patient Global Impression of Improvement (PGI-I) is a patient-reported measure of perceived improvement with treatment, as assessed on a scale of 1 (very much better) to 7 (very much worse). Included here are participants who had improvement as indicated by a rating of 1 (very much better), 2 (much better).
Time Frame: 6 months through 60 Months
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
Number analyzed (Participants) | 116 | 118 | 112
Participants
  06 Months: number analyzed (Participants) | 112 | 114 | 109
  06 Months: Improvement | 96 | 108 | 98
  06 Months: No improvement | 16 | 6 | 11
  12 Months: number analyzed (Participants) | 110 | 108 | 104
  12 Months: Improvement | 101 | 100 | 96
  12 Months: No improvement | 9 | 8 | 8
  24 Months: number analyzed (Participants) | 97 | 95 | 104
  24 Months: Improvement | 87 | 90 | 97
  24 Months: No improvement | 10 | 5 | 7
  36 Months: number analyzed (Participants) | 91 | 93 | 89
  36 Months: Improvement | 79 | 88 | 84
  36 Months: No improvement | 12 | 5 | 5
  48 Months: number analyzed (Participants) | 73 | 72 | 73
  48 Months: Improvement | 58 | 68 | 67
  48 Months: No improvement | 15 | 4 | 6
  60 Months: number analyzed (Participants) | 41 | 37 | 37
  60 Months: Improvement | 33 | 33 | 34
  60 Months: No improvement | 8 | 4 | 3

ADVERSE EVENTS:
Time Frame: 60 Months
Arm/Group | Native Tissue | Sacral Colpopexy | Transvaginal Mesh
All-Cause Mortality (participants affected / at risk) | 2/123 | 1/121 | 5/116
Serious Adverse Events (participants affected / at risk) | 14/123 | 24/121 | 25/116
Other Adverse Events (participants affected / at risk) | 100/123 | 88/121 | 91/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Native Tissue (N=123) | Sacral Colpopexy (N=121) | Transvaginal Mesh (N=116)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Abdominal adhesions (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Colitis microscopic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2)
Constipation (Gastrointestinal disorders) | 2 (3) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Levator syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (4)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 2 (6) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Creutzfeldt-Jakob disease (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bladder injury (Injury, poisoning and procedural complications) | 5 (7) | 5 (6) | 4 (5)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Incision site haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural complication (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) | 0 (0) | 0 (0)
Rectal injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Ureteric injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Gastrointestinal cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Metastasis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
Nerve compression (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (2)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Renal mass (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 3 (3) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0) | 2 (2)
Pelvic haematoma (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bladder neck suspension (Surgical and medical procedures) | 1 (1) | 2 (2) | 0 (0)
Hip arthroplasty (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Hospitalisation (Surgical and medical procedures) | 2 (2) | 1 (1) | 1 (1)
Intra-thoracic aortic aneurysm repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Thyroidectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Vaginal prolapse repair (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Thrombophlebitis (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Native Tissue (N=123) | Sacral Colpopexy (N=121) | Transvaginal Mesh (N=116)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 2 (3)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1) | 1 (1)
Eye swelling (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1)
Abdominal pain lower (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 6 (7) | 10 (11) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2)
Faecal incontinence (Gastrointestinal disorders) | 13 (13) | 9 (9) | 12 (12)
Faecaloma (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal cyst (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Levator syndrome (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0)
Painful defaecation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Proctalgia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Rectal prolapse (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Adhesion (General disorders) | 0 (0) | 1 (1) | 0 (0)
Asthenia (General disorders) | 1 (2) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 2 (2)
Device malfunction (General disorders) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 1 (1) | 0 (0) | 0 (0)
Granuloma (General disorders) | 0 (0) | 1 (1) | 0 (0)
Hypothermia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Medical device site pain (General disorders) | 0 (0) | 1 (1) | 0 (0)
Medical device site reaction (General disorders) | 11 (12) | 5 (6) | 8 (9)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1)
Bile duct stenosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1) | 0 (0) | 0 (0)
Bacterial vaginosis (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Bartholin's abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Cystitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 1 (1) | 1 (1)
Fungal infection (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 2 (2) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 58 (93) | 35 (51) | 60 (93)
Vaginal infection (Infections and infestations) | 5 (6) | 4 (4) | 11 (13)
Vulvitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal mycotic infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Back injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Bladder injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 2 (2)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Incision site pain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Postoperative fever (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (2) | 1 (1)
Procedural vomiting (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 1 (1)
Suture related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Urinary retention postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Vaginal laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
Culture urine (Investigations) | 0 (0) | 0 (0) | 1 (1)
Endoscopy upper gastrointestinal tract (Investigations) | 0 (0) | 0 (0) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Bursitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Coccydynia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 2 (2)
Osteitis deformans (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Vulval cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Neuromyopathy (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0)
Piriformis syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Sciatica (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Bladder dysfunction (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Calculus bladder (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 1 (1) | 2 (2) | 1 (2)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 2 (2)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hydroureter (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertonic bladder (Renal and urinary disorders) | 2 (2) | 1 (1) | 1 (1)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Nocturia (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Obstructive uropathy (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pelvi-ureteric obstruction (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Pollakiuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Stress urinary incontinence (Renal and urinary disorders) | 10 (10) | 22 (22) | 17 (18)
Urethral caruncle (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urge incontinence (Renal and urinary disorders) | 30 (32) | 34 (35) | 24 (27)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 10 (11) | 7 (7) | 13 (16)
Urine flow decreased (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Atrophic vulvovaginitis (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 6 (6)
Bartholin's cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Cystocele (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 0 (0)
Dyspareunia (Reproductive system and breast disorders) | 8 (9) | 6 (6) | 5 (5)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 6 (6) | 8 (8) | 5 (5)
Perineal erythema (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 3 (3)
Vaginal haematoma (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal haemorrhage (Reproductive system and breast disorders) | 7 (7) | 2 (2) | 3 (3)
Vaginal odour (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vaginal perforation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulval disorder (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vulval polyp (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvar erosion (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
Vulvovaginal adhesion (Reproductive system and breast disorders) | 1 (1) | 1 (1) | 1 (1)
Vulvovaginal discomfort (Reproductive system and breast disorders) | 1 (1) | 2 (2) | 3 (3)
Vulvovaginal dryness (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 1 (1)
Vulvovaginal pruritus (Reproductive system and breast disorders) | 2 (2) | 1 (1) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (2)
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Excessive granulation tissue (Skin and subcutaneous tissue disorders) | 16 (16) | 2 (2) | 7 (8)
Lichen sclerosus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Bladder neck suspension (Surgical and medical procedures) | 1 (1) | 3 (3) | 2 (2)
Cataract operation (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (2)
Colporrhaphy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Cystocele repair (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Emergency care (Surgical and medical procedures) | 2 (2) | 0 (0) | 1 (1)
Laparotomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Office visit (Surgical and medical procedures) | 3 (3) | 0 (0) | 1 (1)
Prolapse repair (Surgical and medical procedures) | 1 (1) | 0 (0) | 0 (0)
Stent placement (Surgical and medical procedures) | 0 (0) | 0 (0) | 1 (1)
Surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Urinary incontinence surgery (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Vaginal prolapse repair (Surgical and medical procedures) | 3 (4) | 0 (0) | 0 (0)
Hot flush (Vascular disorders) | 0 (0) | 2 (2) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Thrombophlebitis superficial (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/73/NCT02676973/Prot_000.pdf
  • Statistical Analysis Plan (2023-02-20): https://cdn.clinicaltrials.gov/large-docs/73/NCT02676973/SAP_001.pdf